CLINICAL TRIAL: NCT04800640
Title: Role of Transcutaneous Electrical Nerve Stimulation in Pain Relief and Pulmonary Function in Patients Undergoing Bariatric Surgery
Brief Title: Use of Electroanalgesia in Pain and Pulmonary Function.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11613219.0.0000.5219
Record Dates: First submitted 2020-03-23; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Bariatric Surgery; Obesity, Morbid
Keywords: Spirometry; Electroanalgesia; Bariatric Surgery
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: This is an uncontrolled cross-sectional clinical trial with a sample of 132 individuals between 18 and 50 years of age in a hospital in the West of Paraná. Pain assessment will be performed through analogue pain scale, pulmonary function through spirometry and respiratory muscle strength through manovacuometry. Four TENS applications will be performed for a period of 30 minutes.
Masking Description: He sample will consist of 132 individuals, of both men and women, where they will be randomly included in two groups: 1) Intervention group composed of 66 patients who will effectively receive the treatment through electroanalgesia via TENS; and 2) Control Group, which will also consist of 66 individuals; however, they will not be subjected to electroanalgesia. For division of groups, a sortition will be carried out through envelopes where it will be decided to which study group the patient will be allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Electroanalgesia (No Intervention): The sample will consist of 132 individuals, of both sexes, where they will be randomly included in two groups: 1) Intervention group composed of 66 patients who will effectively receive the treatment through electroanalgesia through TENS; and 2) Control Group, which will also consist of 66 individuals; however, they will not be subjected to electroanalgesia
- Electroanalgesia (Experimental): The sample will consist of 132 individuals, of both sexes, where they will be randomly included in two groups: 1) Intervention group composed of 66 patients who will effectively receive the treatment through electroanalgesia through TENS; and 2) Control Group, which will also consist of 66 individuals; however, they will not be subjected to electroanalgesia
  Interventions: Other: Experimental: Electroanalgesia

INTERVENTIONS:
Other: Experimental: Electroanalgesia — The sample will consist of 66 individuals, of both men and women, where they will be randomly included in two groups: Intervention group composed of 33 patients who will effectively receive the treatment through electroanalgesia via TENS;
  Arms: Electroanalgesia

SUMMARY:
It is a consensus in the literature that changes in lifestyle and carbohydrate-rich diet are part of a context that has led to an obesity pandemic. Its treatment is multidisciplinary, however, in many cases, conventional therapy has no effect, requiring surgical intervention. The latter, in turn, is not free of risks and causes important changes in lung function. Therefore, this study aims to evaluate the effect of electroanalgesia through conventional transcutaneous nerve stimulation (TENS) on pulmonary function in the postoperative period of bariatric surgery.

DETAILED DESCRIPTION:
This is an uncontrolled cross-sectional clinical trial with a sample of 66 individuals between 18 and 50 years of age in a hospital in the West of Paraná. Pain assessment will be performed through analogue pain scale, pulmonary function through spirometry and respiratory muscle strength through manovacuometry. Four TENS applications will be performed for a period of 30 minutes. Through this research, it is expected that the patients who perform TENS present a reduction in postoperative pain and, consequently, a lower impact on lung function.

ELIGIBILITY:
Inclusion Criteria:

* This research will include patients who are in the postoperative period of bariatric surgery and who are aged 18 years or over

Exclusion Criteria:

* Patients over the age of 50;
* Individuals who present hemodynamic instability in the postoperative period;
* Use of mechanical ventilation for more than 24 hours;
* Contraindications regarding the use of TENS (presence of a cardiac pacemaker, hypersensitivity regarding the use of TENS);
* Previous history of epilepsy;
* Pregnant women during the first trimester;
* Patients with a score, on the Glasgow coma scale (Appendix I), less than 15;
* Patients who choose to withdraw during the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
As a primary endpoint, pain using the visual analog pain scale. | 5 days.
  This scale is considered valid to predict the level of pain in the postoperative period of bariatric surgery. The value being zero without pain and ten maximum pain.

SECONDARY OUTCOMES:
Evaluate changes in the strength of respiratory muscles, using manovacuometry. | 5 days.
  The change in manovacuometry can reduce surgical complications.
To evaluate lung function in patients in the postoperative period of bariatric surgery using spirometry. | 5 days.
  The change in lung function can reduce surgical complications.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar A Luchesa, MSc, Principal Investigator — Centro Universitário FAG
Locations (1):
- Centro universitário augusto motta, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benedetti F, Amanzio M, Casadio C, Cavallo A, Cianci R, Giobbe R, Mancuso M, Ruffini E, Maggi G. Control of postoperative pain by transcutaneous electrical nerve stimulation after thoracic operations. Ann Thorac Surg. 1997 Mar;63(3):773-6. doi: 10.1016/s0003-4975(96)01249-0. PMID 9066400
- [Background] Bjordal JM, Johnson MI, Ljunggreen AE. Transcutaneous electrical nerve stimulation (TENS) can reduce postoperative analgesic consumption. A meta-analysis with assessment of optimal treatment parameters for postoperative pain. Eur J Pain. 2003;7(2):181-8. doi: 10.1016/S1090-3801(02)00098-8. PMID 12600800
- [Background] Cipriano G Jr, de Camargo Carvalho AC, Bernardelli GF, Tayar Peres PA. Short-term transcutaneous electrical nerve stimulation after cardiac surgery: effect on pain, pulmonary function and electrical muscle activity. Interact Cardiovasc Thorac Surg. 2008 Aug;7(4):539-43. doi: 10.1510/icvts.2007.168542. Epub 2008 Apr 16. PMID 18417519
- [Background] Erdogan M, Erdogan A, Erbil N, Karakaya HK, Demircan A. Prospective, Randomized, Placebo-controlled Study of the Effect of TENS on postthoracotomy pain and pulmonary function. World J Surg. 2005 Dec;29(12):1563-70. doi: 10.1007/s00268-005-7934-6. PMID 16331341
- [Derived] Luchesa CA, Lopes AJ. Role of Transcutaneous Electric Nerve Stimulation in Pain and Pulmonary Function in Patients after Bariatric Surgery. Rehabil Res Pract. 2022 Jun 2;2022:9138602. doi: 10.1155/2022/9138602. eCollection 2022. PMID 35692935